CLINICAL TRIAL: NCT03126097
Title: A Phase 1, Open-label Study in Healthy Female Subjects to Investigate the Drug-drug Interaction Between JNJ-64155806 and Ethinylestradiol/Drospirenone
Brief Title: A Study to Investigate the Interaction Between JNJ-64155806 and Ethinylestradiol/Drospirenone in Healthy Females
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: Study stopping rules were met.
Sponsor: Janssen Research & Development, LLC (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CR108266; 64155806FLZ1001 (Other: Janssen Research & Development, LLC)
Record Dates: First submitted 2017-04-13; First posted 2017-04-24 (Actual); Last update posted 2017-09-01 (Actual); Status verified 2017-08

CONDITIONS: Healthy
MeSH Terms: interventions — Ethinyl Estradiol; drospirenone

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- JNJ-64155806+COCP+JNJ-64155806 with COCP (Experimental): Participants will receive JNJ-64155806 150 milligram (mg) twice daily (BID) under fed conditions on Days 1 to 7 [JNJ-64155806 Alone Phase] followed by a 10-day washout phase; followed by Ethinylestradiol/drospirenone 0.02 mg/3 mg given as a combined oral contraceptive pill (COCP) once daily (QD) on Days 18 to 41 and COCP placebo QD on Days 42 to 45 [COCP Lead-in Phase]; further followed by COCP QD on Days 46 to 69 (on Days 59 to 66 under fed condition), JNJ-64155806 150 mg BID (under fed conditions) on Days 60 to 66, and COCP placebo QD on Days 70 to 73 [JNJ-64155806 + COCP Co-administration Phase].
  Interventions: Drug: JNJ-64155806 150 mg; Drug: Ethinylestradiol/drospirenone 0.02 mg/3 mg; Drug: COCP Placebo

INTERVENTIONS:
Drug: JNJ-64155806 150 mg — JNJ-64155806 150 mg (3*50 mg tablet) twice daily will be administered under fed conditions on Days 1 to 7 [JNJ-64155806 Alone Phase] and on Days 60 to 66 [JNJ-64155806 + COCP Coadministration Phase].
Drug: Ethinylestradiol/drospirenone 0.02 mg/3 mg — Each tablet contains 3 mg drospirenone and 0.02 mg ethinylestradiol administered as combined oral contraceptive pill (COCP) given on Days 18 to 41 (lead-in phase), Days 46 to 69 (coadministration phase - Days 59 to 66 under fed conditions).
Drug: COCP Placebo — Participant will receive COCP placebo tablets once daily on Days 42 to 45 (lead-in phase) and Days 70 to 73 (JNJ-64155806 + COCP coadministration phase).

SUMMARY:
The primary purpose of this study is to evaluate the effect of single and multiple doses of JNJ-64155806 on the steady-state pharmacokinetics (PK) of ethinylestradiol and drospirenone and vice versa in healthy female participants.

ELIGIBILITY:
Inclusion Criteria:

* Participant must be female of childbearing potential with a normal menstrual cycle, not using oral contraceptives in the 30 days prior to screening
* Participant must have a body mass index (BMI; weight in kilogram (kg) divided by the square of height in meters [m]) of 18.0 to 30.0 kg/m^2, extremes included, and a body weight not less than (<) 50.0 kg
* Participant must be willing and able to adhere to the requirements, instructions, and prohibitions and restrictions specified in this protocol, and is likely to complete the study as planned
* Participant must be healthy on the basis of physical examination, medical history, vital signs, 12-lead electrocardiogram (ECG), and clinical laboratory tests performed at screening. If the results of the biochemistry panel, hematology, or urinalysis are outside the normal reference ranges, the participant may be included only if the investigator judges the abnormalities or deviations from normal to be not clinically significant. This determination must be recorded in the participant's source documents and initialed by the investigator
* Participants must be willing to start ethinylestradiol/drospirenone contraception during the COCP lead-in and JNJ-64155806 + COCP coadministration phases

Exclusion Criteria:

* Participant is a woman who is pregnant as confirmed by a positive beta human chorionic gonadotropin (beta-hCG) laboratory test, or who was pregnant within 6 months prior to study start, or who is breast-feeding, or who is planning to become pregnant from signing of the informed consent form (ICF) until 90 days after the last dose of study drug
* Participant with creatinine clearance of less than (<) 90 milliliter per minute (mL/min) (Chronic Kidney Disease Epidemiology Collaboration [CKD-EPI] equation)
* Participant with a clinically significant cardiovascular, respiratory, renal, gastrointestinal, hematologic, neurologic (syncope or seizures), thyroid, or any other medical illness or psychiatric disorder, as determined by the investigator and/or sponsor's medical monitor
* Participant has any condition for which, in the opinion of the investigator, participation would not be in the best interest of the participant (example, compromise the well-being), or that could prevent, limit, or confound the protocol-specified assessments
* Participant with currently active gynecological disorders including, but not limited to, vaginal bleeding without an obvious reason and hyperprolactinemia with or without galactorrhea

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 18 (Actual)
Dates: Start 2017-04-13 (Actual); Primary Completion 2017-05-26 (Actual); Study Completion 2017-05-26 (Actual)

PRIMARY OUTCOMES:
Trough Plasma Concentration (Ctrough) for Ethinylestradiol | Days 57, 58, 59, 60, 66
  The Ctrough is the plasma concentration before dosing.
Trough Plasma Concentration (Ctrough) for Drospirenone | Days 57, 58, 59, 60, 66
  The Ctrough is the plasma concentration before dosing.
Minimum Observed Plasma Concentration (Cmin) for Ethinylestradiol | Days 59, 60, 66: Predose, 0.5, 1, 2, 3, 4, 6, 8, 12, 16, 20, and 24 hours postdose
  The Cmin is the minimum observed plasma concentration.
Minimum Observed Plasma Concentration (Cmin) for Drospirenone | Days 59, 60, 66: Predose, 0.5, 1, 2, 3, 4, 6, 8, 12, 16, 20, and 24 hours postdose
  The Cmin is the minimum observed plasma concentration.
Maximum Observed Plasma Concentration (Cmax) for Ethinylestradiol | Days 59, 60, 66: Predose, 0.5, 1, 2, 3, 4, 6, 8, 12, 16, 20, and 24 hours postdose
  The Cmax is the maximum observed plasma concentration.
Maximum Observed Plasma Concentration (Cmax) for Drospirenone | Days 59, 60, 66: Predose, 0.5, 1, 2, 3, 4, 6, 8, 12, 16, 20, and 24 hours postdose
  The Cmax is the maximum observed plasma concentration.
Time to Reach Maximum Observed Plasma Concentration (Tmax) for Ethinylestradiol | Days 59, 60, 66: Predose, 0.5, 1, 2, 3, 4, 6, 8, 12, 16, 20, and 24 hours postdose
  The Tmax is defined as actual sampling time to reach maximum observed analyte concentration.
Time to Reach Maximum Observed Plasma Concentration (Tmax) for Drospirenone | Days 59, 60, 66: Predose, 0.5, 1, 2, 3, 4, 6, 8, 12, 16, 20, and 24 hours postdose
  The Tmax is defined as actual sampling time to reach maximum observed analyte concentration.
Average Plasma Concentration (C24h) at 24hours for Ethinylestradiol | Days 59, 60, 66
  C24h is observed analyte concentration at 24 hours.
Average Plasma Concentration (C24h) at 24hours for Drospirenone | Days 59, 60, 66
  C24h is observed analyte concentration at 24 hours.
Average Plasma Concentration (Cavg) for Ethinylestradiol | Days 59, 60, 66
  Cavg is average analyte concentration at steady state, calculated as: AUC24h/24 hours at steady state [24 hours equal to (=) dosing interval].
Average Plasma Concentration (Cavg) for Drospirenone | Days 59, 60, 66
  Cavg is average analyte concentration at steady state, calculated as: AUC24h/24 hours at steady state [24 hours equal to (=) dosing interval].
Area Under the Plasma Concentration-time Curve From Time Zero to 24 Hours (AUC[0-24h]) for Ethinylestradiol | Days 59, 60, 66
  The AUC(0-24h) is the area under the plasma concentration time curve from time zero to 24 hours.
Area Under the Plasma Concentration-time Curve From Time Zero to 24 Hours (AUC[0-24h]) for Drospirenone | Days 59, 60, 66
  The AUC(0-24h) is the area under the plasma concentration time curve from time zero to 24 hours.
Fluctuation Index (FI) for Ethinylestradiol | Days 59, 60, 66
  FI is the percentage fluctuation (variation between maximum and minimum concentration at steady state), calculated as: 100*([Cmax-Cmin]/Cavg).
Fluctuation Index (FI) for Drospirenone | Days 59, 60, 66
  FI is the percentage fluctuation (variation between maximum and minimum concentration at steady state), calculated as: 100*([Cmax-Cmin]/Cavg).
Ratio of Cmin Values Between Test and Reference (Ratio Cmin,test/ref) for Ethinylestradiol | Days 59, 60, 66
  Ratio Cmin,test/ref is the ratio of individual Cmin values between test and reference treatment. Test is Day 60 (JNJ-64155806 single dose + ethinylestradiol/drospirenone) or Day 66 (JNJ-64155806 multiple dose + ethinylestradiol/drospirenone) and Reference is Day 59 (ethinylestradiol/drospirenone alone).
Ratio of Cmin Values Between Test and Reference (Ratio Cmin,test/ref) for Drospirenone | Days 59, 60, 66
  Ratio Cmin,test/ref is the ratio of individual Cmin values between test and reference treatment. Test is Day 60 (JNJ-64155806 single dose + ethinylestradiol/drospirenone) or Day 66 (JNJ-64155806 multiple dose + ethinylestradiol/drospirenone) and Reference is Day 59 (ethinylestradiol/drospirenone alone).
Ratio of Cmax Values Between Test and Reference Treatment (Ratio Cmax,test/ref) for Ethinylestradiol | Days 59, 60, 66
  Ratio Cmax,test/ref is the ratio of individual Cmax values between test and reference treatment. Test is Day 60 (JNJ-64155806 single dose + ethinylestradiol/drospirenone) or Day 66 (JNJ-64155806 multiple dose + ethinylestradiol/drospirenone) and Reference is Day 59 (ethinylestradiol/drospirenone alone).
Ratio of Cmax Values Between Test and Reference Treatment (Ratio Cmax,test/ref) for Drospirenone | Days 59, 60, 66
  Ratio Cmax,test/ref is the ratio of individual Cmax values between test and reference treatment. Test is Day 60 (JNJ-64155806 single dose + ethinylestradiol/drospirenone) or Day 66 (JNJ-64155806 multiple dose + ethinylestradiol/drospirenone) and Reference is Day 59 (ethinylestradiol/drospirenone alone).
Ratio of AUC(0-24h) Values Between Test and Reference (Ratio AUC[0-24h],test/ref) for Ethinylestradiol | Days 59, 60, 66
  Ratio AUC(0-24h),test/ref is the ratio of individual AUC(0-24h) values between test and reference treatment. Test is Day 60 (JNJ-64155806 single dose + ethinylestradiol/drospirenone) or Day 66 (JNJ-64155806 multiple dose + ethinylestradiol/drospirenone) and Reference is Day 59 (ethinylestradiol/drospirenone alone).
Ratio of AUC(0-24h) Values Between Test and Reference Treatment (Ratio AUC[0-24h],test/ref) for Drospirenone | Days 59, 60, 66
  Ratio AUC(0-24h),test/ref is the ratio of individual AUC(0-24h) values between test and reference treatment. Test is Day 60 (JNJ-64155806 single dose + ethinylestradiol/drospirenone) or Day 66 (JNJ-64155806 multiple dose + ethinylestradiol/drospirenone) and Reference is Day 59 (ethinylestradiol/drospirenone alone).

SECONDARY OUTCOMES:
Number of Participants With Adverse Events as a Measure of Safety and Tolerability | From Signing of Informed Consent Form (ICF) till End of Study (Day 73)
  An adverse event is any untoward medical event that occurs in a participant administered an investigational product, and it does not necessarily indicate only events with clear causal relationship with the relevant investigational product.
Minimum Observed Plasma Concentration (Cmin) for JNJ-64155806 | Days 1, 7, 60, 66
  The Cmin is the minimum observed plasma concentration.
Maximum Observed Plasma (Cmax) for JNJ-64155806 | Days 1, 7, 60, 66
  The Cmax is the maximum observed plasma concentration.
Time to Reach Maximum Observed Plasma Concentration (Tmax) for JNJ-64155806 | Days 1, 7, 60, 66
  The Tmax is defined as actual sampling time to reach maximum observed analyte concentration.
Area Under the Plasma Concentration-time Curve From Time Zero to 12 Hours (AUC[0-12h]) for JNJ-64155806 | Days 1, 7, 60, 66
  The AUC(0-12h) is the area under the plasma concentration time curve from time zero to 12 hours.
Area Under the Plasma Concentration-time Curve From 12 Hours to 24 Hours (AUC[12-24h]) for JNJ-64155806 | Days 1, 7, 60, 66
  The AUC(12h-24h) is the area under the plasma concentration time curve from time 12 hours to 24 hours.
Trough Plasma Concentration (Ctrough) for JNJ-64155806 | Days 5, 6, 7, 64, 65, 66
  Ctrough is the plasma concentration before dosing or at the end of the dosing interval of any dose other than the first dose in a multiple dosing regimen.
Average Analyte Concentration (Cavg) for JNJ-64155806 | Days 7 and 66
  Cavg is average analyte concentration at steady state, calculated as: AUC24h/24 hours at steady state [24 hours equal to (=) dosing interval].
Fluctuation Index (FI) for JNJ-64155806 | Days 7 and 66
  FI is the percentage fluctuation (variation between maximum and minimum concentration at steady state).

CONTACTS AND LOCATIONS:
Overall Officials: Janssen Research & Development, LLC Clinical Trial, Study Director — Janssen Research & Development, LLC
Locations (1):
- Celerion, Tempe, Arizona, United States